CLINICAL TRIAL: NCT03741218
Title: Potential Modulatory Effect of Whole Grape on Second-meal Tolerance in Obese Subjects: Role of Polyphenols
Brief Title: Grape Polyphenols and Second-meal Effect
Acronym: GRAPESECOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Jara Pérez-Jiménez, Principal Investigator, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HRG_2018
Record Dates: First submitted 2018-11-13; First posted 2018-11-14 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Obesity
Keywords: Polyphenols; Obesity; Grape; Postprandial; Insulin resistance; Second meal effect
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: GRAP: dried and milled grape pomaces. PLA: control period. All the subjects will pass the two periods: one half will receive the acute PLA supplementation followed by the acute GRAP supplementation, and the other half will do it inversely. The assignment to each order will be done randomly. Both period will be separated by a two weeks washing period.
Who Masked: Participant, Care Provider
Masking Description: GRAP and PLA will have the same aspect, so neither the participant and the care provider will know the received treatment at each stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): All subjects will receive a high-fat breakfast and a medium-fat lunch twice. They will consume together with the breakfast the placebo (PLA) the first time and grape (GRAP) the second time.
  Interventions: Other: Freeze-dried grape (GRAP)/Placebo (PLA)
- 2 (Experimental): All subjects will receive a high-fat breakfast and a medium-fat lunch twice. They will consume together with the breakfast grape (GRAP) the first time and the placebo (PLA) the second time.
  Interventions: Other: Freeze-dried grape (GRAP)/Placebo (PLA)

INTERVENTIONS:
Other: Freeze-dried grape (GRAP)/Placebo (PLA) — The subjects will receive, after overnight fasting, either a monodose of freeze-dried grapes (equivalent to 300 g of fresh grapes) or isocaloric placebo solved in water, together with a high-fat breakfast. Blood samples will be collected before the intake, up to 5 h after breakfast, then a medium-fat lunch will be provided and blood samples will be collected for three additional hours. A total of 10 samples will be collected: 0-30-60-120-180-240-300-330-360-420 min. Both interventions will be separated by two weeks. Subjects will be instructed not to modify their dietary habits during the development of the study, but during the 72 h before each visit they will have to restrict the intake of polyphenol-rich foods (a detailed list will be provided).

SUMMARY:
The aim of this is study is to evaluate the effects of a single intake of grapes (a polyphenol-rich food) in postprandial metabolism in subjects with obesity, including a first intake (high-fat breakfast) after overnight fasting a second one (medium-fat lunch). Studies on the effects of polyphenols on postprandial (glucidic and lipidic) metabolism have commonly been performed in animal models and have used grape extracts, ignoring the whole pool of polyphenols present in grapes (extractable and non-extractable polyphenols). Besides, the contribution of polyphenols to the so-called second-meal effect has not been explored. It should be highlighted that this study aims to explore the potential beneficial role of fresh grapes, consumed as fruit; in order to ensure the stability of the product, they will be provided as freeze-dried milled material, but the amount received by the subjects could be incorporated into a common diet, being equivalent to 300 g of fresh grapes.

DETAILED DESCRIPTION:
Twenty-five subjects with obesity will be were recruited. Detailed inclusion and exclusion criteria are provided below.

The subjects will receive, after overnight fasting, either a monodose of freeze-dried grapes (equivalent to 300 g of fresh grapes) or isocaloric placebo solved in water, together with a high-fat breakfast. Blood samples will be collected before the intake, up to 5 h after breakfast, then a medium-fat lunch will be provided and blood samples will be collected for three additional hours. Both interventions will be separated by two weeks. The following determinations will be performed in blood samples collected at different periods: glucose, insulin, triglycerides, uric acid, viscosity, antioxidant capacity. Additionally, a satiety test will be provided. It is expected that grape supplementation, as compared with an isocaloric placebo, causes significant modifications in all the parameters indicated. Nevertheless, the primary outcome of this study is the area under the curve for glucose after the second meal (300-420 min from basal time).

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI = 30-40 kg/m2).

Exclusion Criteria:

* Subjects with a pharmaceutical treatment set to modify blood pressure, lipid profile or glucose.
* Subjects with diagnoses of type 2 diabetes, cardiovascular diseases or thyroid diseases.
* Values above the following ones: glucose, > 115 mg/dL; triglycerides, > 350 mg/dL; total cholesterol, > 280 mg/dL; systolic blood pressure, > 150 mmHg; diastolic blood pressure, > 100 mmHg
* Previous bariatric surgery.
* Volunteers participating in other studies (currently or during last year) or weight loss plans.
* Pregnant or breastfeeding women.
* Adherence to vegetarian diets or usual consumption of dietary supplements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose (300-420 min) | Up to two months
  Changes of postprandial blood glucose as result of supplementation with grapes, measured area under the curve for the period 300-420 min

OTHER OUTCOMES:
Postprandial glucose and insulin | Up to four months
  Changes of blood glucose (0-320 min) and insulin (0-300 and 300-420 min) as result of supplementation with grapes
Plasma triglycerides | Up to four months
  Changes of plasma triglycerides (0-300 and 300-420 min) as result of supplementation with grapes
Plasma uric acid | Up to four months
  Changes of plasma uric acid (0-300 and 300-420 min) as result of supplementation with grapes
Plasma antioxidant capacity | Up to five months
  Changes of plasma antioxidant capacity (0-300 and 300-420 min) as result of supplementation with grapes
Plasma viscosity | Up to six months
  Changes of plasma viscosity (0-300 and 300-420 min) as result of supplementation with grapes.
Satiety | Up to three months
  Changes of satiety (0-300 and 300-420 min) as result of supplementation with grapes.

CONTACTS AND LOCATIONS:
Overall Officials: Jara Pérez-Jiménez, PhD, Principal Investigator — Institute of Food Science, Technology and Nutrition (ICTAN-CSIC)
Locations (1):
- Institute of Food Science, Technology and Nutrition, National Research Council (ICTAN-CSIC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Diez E, Cuesta-Hervas M, Veses-Alcobendas AM, Alonso-Gordo O, Garcia-Maldonado E, Martinez-Suarez M, Herranz B, Vaquero MP, Alvarez MD, Perez-Jimenez J. Acute supplementation with grapes in obese subjects did not affect postprandial metabolism: a randomized, double-blind, crossover clinical trial. Eur J Nutr. 2021 Aug;60(5):2671-2681. doi: 10.1007/s00394-020-02451-6. Epub 2021 Jan 2. PMID 33386890